CLINICAL TRIAL: NCT00860743
Title: Respiratory and Autonomic Plasticity Following Intermittent Hypoxia
Acronym: RAP-IH
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: PULM-014-08F; GRANT00507547 (Other Grant/Funding Number: VA Merit)
Record Dates: First submitted 2009-03-10; First posted 2009-03-12 (Estimated); Results first posted 2015-02-25 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-09

CONDITIONS: Sleep Apnea Syndromes
Keywords: intermittent hypoxia; ventilatory long-term facilitation; autonomic nervous system plasticity
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (No Intervention): We plan to study 10 males and 10 females with moderate obstructive sleep apnea (OSA), and 10 healthy males and 10 healthy females. The males and the females will be matched based on age, race, sex and body mass index. The OSA and control participants will be exposed to intermittent hypoxia and "sham" intermittent hypoxia during wakefulness and sleep.
- ANTIOXIDANT COCKTAIL (Experimental): We plan to study 10 male participants with moderate obstructive sleep apnea (OSA) and 10 male control participants matched for age, race and body mass index. The OSA and control participants will be exposed to intermittent hypoxia during wakefulness and sleep following administration of an antioxidant or a placebo cocktail that will be presented in a randomized fashion.
  Interventions: Drug: Antioxidant cocktail

INTERVENTIONS:
Drug: Antioxidant cocktail — 120 mg of Coenzyme Q10 (orally), 800 mg of Superoxide Dismutase (orally), 400 IU of Vitamin E (orally) before exposure to intermittent hypoxia. Two doses of 1 g of Vitamin C in 50 cc of saline IV (in the vein) before and after exposure to intermittent hypoxia.
  Arms: ANTIOXIDANT COCKTAIL

SUMMARY:
The prevalence of obstructive sleep apnea is high in the Veteran population. If not treated promptly, sleep apnea may result in daytime fatigue which may lead to increased prevalence of accidents while driving or in the workplace. Recent large scale epidemiological studies have shown that the prevalence of excessive daytime sleepiness increases in individuals who suffer from obstructive sleep apnea. Obstructive sleep apnea may also result in the development of hypertension and other cardiovascular disorders. Previous findings have shown that subjects with sleep apnea have a greater risk for developing coronary vascular disease compared to individuals that do not suffer from sleep apnea Thus, a significant amount of evidence suggests that sleep apnea is a major health concern in the Veteran population. Consequently, determining the mechanisms that may impact on the severity of sleep apnea and increase the prevalence of cardiovascular incidents associated with this disorder is important, as is discovering novel treatments.

DETAILED DESCRIPTION:
Approximately 8 % of the Veteran population in the United States suffers from sleep apnea. Consequences of untreated sleep apnea include increased daytime fatigue, hypertension and stroke. Thus, sleep apnea is a major health concern. One of the primary hallmarks of sleep apnea is exposure to intermittent hypoxia (IH) which occurs as a consequence of central or obstructive apneas. Exposure to IH may lead to neural plasticity (i.e. a change in system performance based on prior experience) of the respiratory and autonomic nervous system. One adaptation that has been shown to manifest itself in animals following exposure to IH is long-term facilitation (LTF) of ventilation and sympathetic nervous system activity (SNSA). This phenomenon is characterized by a gradual increase in respiratory motor activity and SNSA during successive periods of normoxia that separate hypoxic episodes and by activity that persists above baseline levels for up to 90 minutes following exposure to IH. Although LTF of minute ventilation has been well established in animals it has not been observed consistently in healthy humans or in individuals with obstructive sleep apnea. Similarly, although a few studies have shown that exposure to IH leads to increases in SNSA in healthy individuals the magnitude of the response has varied significantly. Findings from animal studies suggest that the manifestation of LTF in humans might in part be dependent on a variety of factors, including prior exposure to IH, arousal state (wake vs. sleep) and gender. Thus, the initial aim of our proposal will establish whether LTF can be induced in healthy humans and individuals with obstructive sleep apnea and whether the magnitude of the response is dependent on those factors mentioned above. Moreover, the initial aim will explore whether the presence of LTF of minute ventilation promotes or mitigates apnea severity. Animal studies have also indicated that LTF of respiratory and autonomic activity may in part be induced by increases in oxidative stress. Thus, the second objective of our proposal will explore whether administration of an antioxidant cocktail impacts respiratory and autonomic nervous system plasticity during wakefulness and sleep following IH. Likewise, the second aim will explore whether administration of an antioxidant cocktail alters apnea severity following exposure to IH. Establishing whether LTF of minute ventilation exists in individuals with sleep apnea is important since activation of this phenomenon could impact on apnea severity across the night. Similarly, LTF of SNSA activity and possibly long-term depression (LTD) of parasympathetic nervous system activity (PNSA) could ultimately lead to persistent increases in blood pressure and heart rate. Furthermore, given that exposure to IH may lead to long-term plasticity of respiratory and autonomic activity that are physiologically detrimental, exploring mechanisms that ultimately lead to treatments that may mitigate or prevent the manifestation of this phenomenon are important.

ELIGIBILITY:
Inclusion Criteria:

Characteristics of OSA subject population:

* Body mass index < 30 kg/m2.
* 20 to 40 years old.
* Newly diagnosed never-treated mild to moderate sleep apnea (i.e. 50 > apnea/hypopnea index >10 events per hour - average nocturnal oxygen saturation > 90%).
* Not pregnant.
* Free of any other known medical conditions.
* Not taking any medication.
* Non-smokers with normal lung function.
* Minimal alcohol consumption (i.e. no more than the equivalent of a glass of wine/day).

Characteristics of control group population:

* Body mass index < 30 kg/m2.
* 20 to 40 years old.
* Apnea/hypopnea index < 5 events per hour.
* Not pregnant.
* Free of any known medical conditions.
* Not taking any medication.
* Non-smokers with normal lung function.
* Minimal alcohol consumption (i.e. no more than the equivalent of a glass of wine/day).

Exclusion Criteria:

* Anything not in inclusion criteria.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2009-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason H Mateika, PhD MS BS, Principal Investigator — John D. Dingell VA Medical Center, Detroit
Locations (1):
- John D. Dingell VA Medical Center, Detroit, Detroit, Michigan, United States

REFERENCES:
- [Result] Mateika JH, Syed Z. Intermittent hypoxia, respiratory plasticity and sleep apnea in humans: present knowledge and future investigations. Respir Physiol Neurobiol. 2013 Sep 15;188(3):289-300. doi: 10.1016/j.resp.2013.04.010. Epub 2013 Apr 12. PMID 23587570
- [Result] Syed Z, Lin HS, Mateika JH. The impact of arousal state, sex, and sleep apnea on the magnitude of progressive augmentation and ventilatory long-term facilitation. J Appl Physiol (1985). 2013 Jan 1;114(1):52-65. doi: 10.1152/japplphysiol.00985.2012. Epub 2012 Nov 8. PMID 23139361

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study recruited participants between the years 2009-2013. The study was completed at the John D. Dingell VA Medical Center.
Pre-assignment Details: 1. Participants did not meet the inclusion criteria. This was typically due to EKG abnormalities or high blood pressure.
  2. Participants completed a "practice run" following consent to introduce them to equipment and procedures. Some participants choose not to continue following the practice run usually because of discomfort.
Groups:
- OSA/Healthy - Males/Females - Wake/Sleep: We plan to study 10 males and 10 females with moderate obstructive sleep apnea (OSA), and 10 healthy males and 10 healthy females. The males and the females will be matched based on age, race, sex and body mass index. The OSA and control participants will be exposed to intermittent hypoxia and "sham" intermittent hypoxia during wakefulness and sleep.
- Arm 2: We plan to study 10 male participants with moderate obstructive sleep apnea (OSA) and 10 male control participants matched for age, race and body mass index. The OSA and control participants will be exposed to intermittent hypoxia during wakefulness and sleep following administration of an antioxidant or a placebo cocktail that will be presented in a randomized fashion.
  Antioxidant cocktail: 120 mg of Coenzyme Q10 (orally), 800 mg of Superoxide Dismutase (orally), 400 IU of Vitamin E (orally) before exposure to intermittent hypoxia. Two doses of 1 g of Vitamin C in 50 cc of saline IV (in the vein) before and after exposure to intermittent hypoxia.
Period: Overall Study
Arm/Group | OSA/Healthy - Males/Females - Wake/Sleep | Arm 2
Started | 40 | 23
Completed | 37 | 23
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Population: Overall 40 participants were enrolled in Aim 1. One OSA male and two healthy male participants were enrolled but withdrew from the study. Thus, the total number that completed Aim 1 was 37 participants.
Groups:
- Aim 1 - OSA Male - Sleep/Wake - Hypoxia/Sham: We plan to study 10 OSA males. These males will be matched with 10 females with moderate obstructive sleep apnea (OSA), 10 healthy males and 10 healthy females. The males and the females will be matched based on age, race, sex and body mass index. The OSA and control participants will be exposed to intermittent hypoxia and "sham" intermittent hypoxia during wakefulness and sleep.
- Aim 1 - OSA Female- Sleep/Wake - Hypoxia/Sham: We plan to study 10 OSA females. These females will be matched with 10 males with moderate obstructive sleep apnea (OSA), 10 healthy males and 10 healthy females. The males and the females will be matched based on age, race, sex and body mass index. The OSA and control participants will be exposed to intermittent hypoxia and "sham" intermittent hypoxia during wakefulness and sleep.
- Aim 1 - Healthy Males- Sleep/Wake - Hypoxia/Sham: We plan to study 10 healthy males. These males will be matched with 10 OSA males and 10 OSA females with moderate obstructive sleep apnea (OSA), and 10 healthy males and 10 healthy females. The males and the females will be matched based on age, race, sex and body mass index. The OSA and control participants will be exposed to intermittent hypoxia and "sham" intermittent hypoxia during wakefulness and sleep.
- Aim 1 - Healthy Females- Sleep/Wake - Hypoxia/Sham: We plan to study 10 males and 10 females with moderate obstructive sleep apnea (OSA), and 10 healthy males and 10 healthy females. The males and the females will be matched based on age, race, sex and body mass index. The OSA and control participants will be exposed to intermittent hypoxia and "sham" intermittent hypoxia during wakefulness and sleep.
- Aim 2 - OSA - Hypoxia - Antioxidant/Placebo: We plan to study 10 male participants with moderate obstructive sleep apnea (OSA) and 10 male control participants matched for age, race and body mass index. The OSA and control participants will be exposed to intermittent hypoxia during wakefulness following administration of an antioxidant or a placebo cocktail that will be presented in a randomized fashion.
  Antioxidant cocktail: 120 mg of Coenzyme Q10 (orally), 800 mg of Superoxide Dismutase (orally), 400 IU of Vitamin E (orally) before exposure to intermittent hypoxia. Two doses of 1 g of Vitamin C in 50 cc of saline IV (in the vein) before and after exposure to intermittent hypoxia.
- Aim 2 - Healthy - Hypoxia - Antioxidant/Placebo: We plan to study 10 male participants with moderate obstructive sleep apnea (OSA) and 10 male control participants matched for age, race and body mass index. The OSA and control participants will be exposed to intermittent hypoxia during wakefulness following administration of an antioxidant or a placebo cocktail that will be presented in a randomized fashion.
- Total: Total of all reporting groups
Arm/Group | Aim 1 - OSA Male - Sleep/Wake - Hypoxia/Sham | Aim 1 - OSA Female- Sleep/Wake - Hypoxia/Sham | Aim 1 - Healthy Males- Sleep/Wake - Hypoxia/Sham | Aim 1 - Healthy Females- Sleep/Wake - Hypoxia/Sham | Aim 2 - OSA - Hypoxia - Antioxidant/Placebo | Aim 2 - Healthy - Hypoxia - Antioxidant/Placebo | Total
Number analyzed (Participants) | 11 | 7 | 12 | 10 | 13 | 10 | 63
Age, Customized [Mean (Standard Deviation); unit: years] | 24.8 (3.1) | 26.6 (5.9) | 25.2 (4.0) | 24.8 (4.1) | 31.2 (6.2) | 29.1 (5.1) | 26.6 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 7 | 0 | 10 | 0 | 0 | 17
  Male | 11 | 0 | 12 | 0 | 13 | 10 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 11 | 7 | 12 | 10 | 13 | 9 | 62
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 5 | 5 | 5 | 4 | 6 | 30
  White | 6 | 2 | 7 | 5 | 9 | 4 | 33
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 7 | 12 | 10 | 13 | 10 | 63

OUTCOME MEASURES:

1. Primary Outcome: Ventilation (Aim 1)
Description: Ventilation was measured before and after exposure to intermittent hypoxia in males and females. Ventilation was measured using a pneumotachograph, which is a flow measuring device.
Time Frame: Within the same experimental session
Measure: Mean (Standard Error); unit: fraction of baseline
Arm/Group | OSA/HEALTHY - MALES/FEMALES - WAKE/SLEEP
Number analyzed (Participants) | 37
fraction of baseline
  OSA male during wakefulness | 1.19 (0.03)
  OSA male during sleep | 1.14 (0.03)
  OSA female during wakefulness | 1.35 (0.03)
  OSA female during sleep | 1.16 (0.05)
  Healthy male during wakefulness | 1.19 (0.03)
  Healthy male during sleep | 1.09 (0.03)
  Healthy female during wakefulness | 1.26 (0.06)
  Healthy female during sleep | 1.08 (0.04)
Statistical Analysis 1: Comparison: OSA/HEALTHY - MALES/FEMALES - WAKE/SLEEP; Test type: Superiority or Other; p = 0.001, ANOVA — P values less than 0.05 are considered statistically significant in this study

2. Primary Outcome: Heart Rate Variability (Aim 2)
Description: Heart rate variability (HRV) was measured before and after exposure to intermittent hypoxia following administration of a placebo or antioxidant cocktail. Heart rate variability refers to beat-to-beat alterations in heart rate. Under resting conditions, the electrocardiogram of healthy individuals reveals periodic variation in R-R intervals. To measure HRV, R-R interval data are presented in a graph, in which the y-axis plots the R-R intervals (ms2), and the x-axis the total number of beats. Spectral analysis of the graph transforms the signal from time to frequency on the x-axis (Hz), by representing the signal as a combination of sine and cosine waves, with different amplitudes and frequencies. The approach uses Fourier transforms. The heart rate spectrum contains a high frequency (0.15-0.4 Hz) component, which is synchronous with respiration and a low frequency (0.04 to 0.15 Hz) component that appears to be mediated by both the vagus and cardiac sympathetic nerves.
Time Frame: Within the same experimental session
Population: Measurements were made before and after intermittent hypoxia following administration of a placebo or antioxidant cocktail. Please note that analysis of the heart rate variability measures for the healthy group have not been completed to date.
Measure: Mean (Standard Error); unit: ms2/Hz
Groups:
- OSA/HEALTHY - HYPOXIA - ANTIOXIDANT/PLACEBO: We plan to study 10 male participants with moderate obstructive sleep apnea (OSA) and 10 male control participants matched for age, race and body mass index. The OSA and control participants will be exposed to intermittent hypoxia during wakefulness and sleep following administration of an antioxidant or a placebo cocktail that will be presented in a randomized fashion.
  Antioxidant cocktail: 120 mg of Coenzyme Q10 (orally), 800 mg of Superoxide Dismutase (orally), 400 IU of Vitamin E (orally) before exposure to intermittent hypoxia. Two doses of 1 g of Vitamin C in 50 cc of saline IV (in the vein) before and after exposure to intermittent hypoxia.
Arm/Group | OSA/HEALTHY - HYPOXIA - ANTIOXIDANT/PLACEBO
Number analyzed (Participants) | 13
ms2/Hz
  OSA before intermittent hypoxia placebo (HF) | 3766.1 (1129.859)
  OSA after intermittent hypoxia placebo (HF) | 2944.9 (935.0)
  OSA before intermittent hypoxia antioxidant (HF) | 3810.5 (1712.2)
  OSA after intermittent hypoxia antioxidant (HF) | 2516.3 (835.8)
  OSA before intermittent hypoxia placebo (LF) | 2737.7 (573.1)
  OSA after intermittent hypoxia placebo (LF) | 2289.1 (568.1)
  OSA before intermittent hypoxia antioxidant (LF) | 2761.6 (629.1)
  OSA after intermittent hypoxia antioxidant (LF) | 1889.9 (336.3)
Statistical Analysis 1: Comparison: OSA/HEALTHY - HYPOXIA - ANTIOXIDANT/PLACEBO; Test type: Superiority or Other; p = 0.2, ANOVA

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/23
Other Adverse Events (participants affected / at risk) | 0/40 | 0/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=40) | Arm 2 (N=23)
premature ventricular contraction (Cardiac disorders) | 0 | 0 — 119 individuals were screened in order to enroll 63 participants in our study. During screening participants were exposed to two episodes of hypoxia. Premature ventricular contractions were recorded from one participant not enrolled in the study.

LIMITATIONS AND CAVEATS:
The primary limitation of this trial was the number of participants that required screening to recruit the participants that met the inclusion criteria for the study. However, once the participants were recruited few withdrew.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes